# Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and

# Vomiting During Pregnancy (A Randomized Control Trial)

تأثير تنفيذ إرشادات "أتاوا" الغذائية على مسار الغثيان والقيئ أثناء الحمل (دراسة تجريبية عشوائية)

By

Noura Mohamed El-toukhi

(M.Sc. Nursing)

Dissertation proposal

Submitted in Partial Fulfillment of the Requirements of the

Doctorate Degree in Midwifery Nursing

#### **Advisors**

Dr. Yousria El-sayed

Professor of Maternal & Newborn Health

Dr. Abeer Saad Zaghloul

Professor of Maternal & Newborn Health

Nursing

Faculty of Nursing

Cairo University

Nursing

Faculty of Nursing -

Cairo University

125 / /2 Ass

Dr. Tamer Mahmoud Assar

Assistant Professor of Obstetrics & Gynacology

Faculty of Medicine

**Benha University** 

J 6.0-9-4

**Faculty of Nursing** 

Cairo University

2020-2021

Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial)

تأثير تنفيذ إر شادات "أتاوا " الغذائية على مسار الغثيان والقيئ أثناء الحمل (دراسة تجربيية عشوانية)

#### Introduction

Nausea and vomiting of pregnancy (NVP) is the most prevalent medical condition associated with pregnancy, affecting up to 80% of pregnant women(Mitsuda, Eitoku, Maeda, Fujieda, & Suganuma, 2019), (Matthews, Haas, O'Mathúna, & Dowswell, 2015). Nausea and vomiting of pregnancy commonly occurs between 5 and 18 weeks of pregnancy. Between 50 and 90% of women with normal pregnancies have some degree of nausea, with or without vomiting. The etiology of NVP is unknown, and symptoms range in severity from mild nausea to the most severe form of vomiting, known as hyperemesis gravidarum (HG). This occurs in 0.3–3.6% of pregnancies, and can potentially result in metabolic disturbances, including dehydration and ketosis (Boelig, Barton, Saccone, Kelly, Edwards, &Berghella, 2018).

There is a relationship between (NVP) during pregnancy and some pregnancy complications as significant relationship with preterm labor (P=0.002), hypertension (P=0.003), anemia (P=0.002), and cesarean section (P=0.009). (Mohamadi, Garkaz, Abolhassani, &BolbolHaghighi, 2020).

Nausea and vomiting of pregnancy often develops by 5<sup>th</sup> to 6<sup>th</sup> weeks of pregnancy and affects 84% of women. The symptoms are usually worst around nine weeks and typically improve by 16 to 18 weeks of pregnancy. However, symptoms continue into the third trimester in 15% to 20% of women and until delivery in 5% of women. (Hassan et al., 2017)

Mild pregnancy-related nausea and vomiting is typically characterized as a pregnant woman feeling nauseated each day and possibly vomiting once or twice/day. (Hinkle, et al, 2016). It is usually not harmful to the fetus, although obviously vomiting daily has a serious impact on a woman's life (ACOG, 2018).

The moderate form of (NVP) is diagnosed when the women's score of Pregnancy Unique Quantification of Emesis and Nausea (PUQE 24) is from 7-12. In one meta-analysis, the odds of miscarriage in women with nausea and vomiting in the first 20 weeks of pregnancy was odds ratio (OR) 0.36 (95% CI 0.2-0.42). The analysis did not correlate outcome with respect to the severity of the disorder, most of the women in the studies had mild symptoms rather than hyperemesis (Hinkle et al, 2016).

Nausea and vomiting of pregnancy is most likely a multifactorial condition and has been associated with many risk factors. Multiple nutrient deficiencies have been identified in association with nausea and vomiting. Women with nausea and vomiting are more likely to be younger, primiparous, female infant sex, twins or triples, history of nausea or vomiting, history of being susceptible to motion sickness, family history of nausea during pregnancy, and less likely to drink alcohol (Roseboom, Ravelli, & Painter, 2011).

د/تامر کھر

Nausea and vomiting of pregnancy was significantly associated with several characteristics, including daily life functioning, quality of life and willingness to become pregnant again. The negative impact was greater the more severe the symptoms were, although considerable adverse effects were also seen among women with mild and moderate NVP symptoms. Women with severe NVP considered terminating the

pregnancy due to NVP, and others considered not to get pregnant again. Severity of NVP remained significantly associated with reduced global quality of life when adjusting for maternal characteristics and illnesses with  $\beta$  (95% CI) = -10.9 (-16.9, -4.9) for severe versus mild NVP (Heitmann, Nordeng, Havnen, Solheimsnes, &Holst, 2017). Nausea and vomiting of pregnancy can also impact women's ability to carry out daily parenting or work tasks. Up to 35% of women with NVP report depression (Bustos, Venkataramanan, & Caritis, 2017).

Treatment and management of NVP depend on severity of symptoms. Time of treatment is of great significance, as early treatment can reduce the severity and intensity of NVP symptoms, decrease the need for hospitalization, reduce time waste for working pregnant women, and diminish psychological disorders and psychiatric problems. However, more evidence is needed to support early intervention. (Davis, 2004).

Nausea and vomiting during pregnancy may be undertreated due to the concerns about the safety of medications however; this does not mean that women do not seek other treatments. It can be more difficult to control symptoms once nausea and vomiting of pregnancy progresses. According to American College of Obstetrics and Gynecology (2018), Treatment in the early stages of NVP can avert more serious complications. Mild to moderate cases can be resolved with changes to lifestyle and diet

Non-pharmacological remedies such as dietary modifications, dehydration prevention, rest, exercise, fresh air breathing, herbal remedies (such as ginger and peppermint), aromatherapy, sleep pattern adjustments, psychotherapy, hypnosis, homeopathy, music therapy, and acupuncture (e.g., electro-accu-puncture, electrical nerve stimulation through the skin, and acupressure), (Boelig, Barton, Saccone, Kelly, Edwards, & Berghella, 2018). Nutritional care and lifestyle changes are important parts of treatment

for NVP. Nutritional modifications, such as use of carbohydrates and carbonated drinks, as well as relaxation techniques are effective in this area. Previous research on women with NVP shows that dietary changes lead to a moderate decline in the symptoms. Also, a recent study showed that women on a high-protein diet experience less severe NVP (Matthews, Haas, Mathúna, &Dowswell, 2015).

Other recommendations for women with NVP include minimizing the time for preparing food, lying down after digestion, eating food in quiet and comfortable places, avoiding warm places with thick odors, drinking liquid half an hour before and after a meal, drinking a cup of herbal tea with honey (such as mint and chamomile), and wearing comfortable clothes. Brushing the teeth after a meal, drinking mint tea, or sucking on peppermint candy after meals can also improve postprandial nausea (ACOG, 2018). However, these recommendations haven't been tested

According to Ottawa guidelines the management of NVP is combination of different regimen recommendations about lifestyle modifications, nutritional therapies, complementary medicine, and acupressure, aims to restore optimal nutrition and quality of life during pregnancy. In addition to general information it includes risk factors, general guidelines, nutritional considerations, suggested foods, and sample menu designed to control nausea and vomiting during pregnancy. The guidelines include no drugs and are based on life style modification and self administered management.

The potential of pharmacologic and non-pharmacologic treatment options have not been studied fully and available evidence is generally of low quality. This negatively affects the quality of patient care There is no evidence to support the effectiveness of dietary restrictions to relieve symptoms, (Matthews 2014).

In Egypt, documented data about prevalence of nausea and vomiting during pregnancy is scares. This is because nausea and vomiting during pregnancy (NVP) are not as a pathological condition to be admitted to the hospital. Therefore, Research has been focusing more on hyperemesis gravidarum (HG) admitted to hospitals. (Mahmoud, 2012)

# Significance of the study

The Ottawa nutritional guidelines are designed by Ottawa Hospital, Canada 2017 for the management of NVP and raising pregnant women's awareness of self-care in order to improve their quality of life. The guideline aims to provide evidence-based instructions for the early treatment of NVP and suggests strategies for the early diagnosis and treatment of this condition in order to prevent hyperemesis gravidarum that need for injection therapy, and increased cost of hospitalization. A study to explore thoughts and attitudes among Norwegian pregnant women and care provider on treatment of NVP and pregnancy care showed that the health care provider perceive NVP as normal so it made the women feel that their distress due to NVP was trivialized by them, and both the care provider and the women showed a reluctant attitude to medical treatment of NVP. The care provider gave the impression of considering medical treatment only after progression of symptoms to becoming quite severe. (Heitmann, Svendsen, Sporsheim, & Holst; 2016).

دا تامر قصر

#### Aim of the Study

To study the impact of applying Ottawa nutritional guidelines on the progress of the course of nausea and vomiting during pregnancy



Conceptual Framework

# Research Hypothesis

Hypothesis: 1

Pregnant women with nausea and vomiting who will follow the Ottawa nutritional guidelines will show improved nausea and vomiting as scored by the modified 24-hour pregnancy-unique quantification of emesis and nausea (PUQE 24) compared to those who receive routine antenatal protocol.

# Subjects and Methods

respet/s

Research Design. Randomized controlled trail (single blind)

is a type of scientific experiment that aims to reduce certain sources of bias when testing the effectiveness of new treatments; this is accomplished by randomly allocating subjects to two or more groups, treating them differently, and then comparing them with respect to a measured response. One group (the experimental group) receives the intervention being assessed, while the other usually called the (control group) receives an alternative treatment, such as a placebo or no intervention. The current study includes two groups (Study group), which will receive routine antenatal care in addition to the Ottawa nutritional guidelines, and (control group), which will receive only routine antenatal care.

# Setting

Antenatal clinic at El: Zahra center will be the setting for collecting the data needed to conduct this study. El: Zahra center a nongovernmental obstetric center affiliated by the Egyptian ministry of health, located in Moshtohor, Toukh, Qualubia governorate, it is equipped to manage primary and referral cases, it provides antenatal care to low risk pregnant women, as well as vaginal deliveries, cesarean section, management of intrapartum complications, early postpartum care, management of postpartum complications in addition to different obstetric and gynecological services as IUD insertion or removal, infertility management, and family planning services. Approximately annually admissions according to its local statistics for the year (5000 case, 2019).

Sample A total of (60) pregnant women who complain of mild to moderate nausea and vomiting, (having a score of 7-12 on the (PUQE 24) will be recruited for this study via simple sampling, subjects who will meet the inclusion criteria will be randomly allocated to either intervention or control groups (N=30) each using sealed opaque envelops. Subjects will be recruited according to the following inclusion criteria: 1) primigravida; 2) gestational age of 7-13 weeks; 3) singleton pregnancy; 4) having a score of 7-12 on the (PUQE 24); 5) can read and write; 6) having phone number; 7) not receiving medications for reducing NVP, except for vitamin B6; 8) wanted pregnancy.

Jes > 1/2

The exclusion criteria will be as follows: 1) subject's unwillingness to continue the study, 2) occurrence of obstetric complications during the study, 3) hyper-emesis gravidarum, 4) having physical or mental disorders; 5) having oral/speech impairments; 6) having assisted reproductive techniques for the present pregnancy; 7) having two consecutive miscarriages before the current pregnancy; 8) old primigravida 9) narcotic use or alcohol drinking, and subjects who will show signs and symptoms of hyperemesis gravidarum during the study will be dropped out and referred to medical care.

Sample size is calculated according to this equation:  $n = \frac{N}{1 + N(e)2}$ , n=sample size, N=population size, e=Co-efficient factor (error),  $n = \frac{70}{1 + 70X0.005} = \frac{70}{1.175} = 60$  Subjects (30) for each group.

#### Randomization

The researcher will attend the study setting to collect the required sample, women who met the eligibility criteria will be numbered by the researcher & randomly every odd number will be recruited in the study, a random assignment and allocation of the participants in each group through using closed opaque envelopes containing card written on it P6 acupressure or control group will be done.

#### **Tools for Data collection**

Required data will be collected by using the following tools:

respetto

<u>1-Structred interview questionnaire Schedule</u> It will be designed by the investigator and will encompasses of a) socio-demographic characteristics of pregnant women, b) history of current pregnancy such as gestational age, gravidity, parity, Ob code, c) data related to history of nausea and vomiting during previous and current

Effect of Implementing Ottawa Guidelines on the Course of Nausea and Vomiting pregnancy. This tool will be designed by the research investigator and approved by panel experts in gynecology and maternity nursing.

2- Modified 24-hour Pregnancy-Unique Quantification of Emesis and nausea (PUQE 24): Quantification of Emesis/Nausea (PUQE 24) Index It is an objective and validated index adopted from (Ebrahimi et al., 2009) and used to measure the severity of symptoms of nausea and vomiting of pregnancy (NVP) in the previous 24 hours. This index contains three questions regarding the length of nausea per day in hours, the number of daily vomiting episodes, and the number of retching episodes. Each PUQE 24 question has a rating from one to five.

Scoring The three (PUQE 24) questions each have a rating from 1–5, thus the composite sum (PUQE 24 score) ranged from 3–15. A score between 3–6 points was defined as mild NVP, 7–12 points as moderate NVP and scores 13 points was classified as severe NVP/HG, in line with former studies.

3-Ottawa nutritional guidelines to help control nausea and vomiting during pregnancy. This guideline aims to provide evidence-based instructions for the early treatment of NVP and suggests strategies for the early diagnosis and treatment of this condition in order to prevent hyperemesis gravidarum, need for injection therapy, and increased cost of hospitalization. Developed by Ottawa Hospital, Canada 2017. This guideline will be used as a guide for intervention and follow up. It includes recommendations about lifestyle modifications, nutritional therapies, complementary medicine, and acupressure.

# Validity and reliability of the tools Structred interview questionnaire Schedule

Tools will be submitted to a panel of three nursing experts in the field of obstetrics and to test the content validity will be carried out according to the panel judgment on clarity of sentences and the appropriateness of content. Internal consistency by Cronbach's  $\alpha$ .

د/ کا فر کھر

The version of PUQE 24-24, is valid as a clinical tool to distinguish between regular

morning sickness and severe nausea and vomiting of pregnancy (Lacasse, Rey, Ferreira,

Morin & Bérard, 2008).

Pilot study

A pilot study will be conducted of 10 % of the sample to test the feasibility of

data collection as, clarity and objectivity of the tools.

**Ethical consideration** 

An official permission to conduct the study will be obtained from the ethical

committee from faculty of nursing Cairo University. Also, an official permission was

granted from the director of setting. The research investigator will introduce her to the

women who met the inclusion criteria and informed them about the aim of the study in

order to obtain their acceptance. All women will be informed that participation in this

study is voluntary; and they can withdraw at any time during the study without giving

reasons and their withdrawal will not affect the care they will receive. An informed

written consent will be obtained from study participants.

**Procedure** 

All registered pregnant women who complain of nausea and vomiting will be invited to

participate in the study. Those who meet the inclusion criteria will be enrolled. The aim

of the study will be explained to subjects to gain their acceptance to participate in the

study, after obtaining the written consent forms, subjects will then be randomly allocated

to either intervention (N=30) or control (N=30) using closed envelopes containing card

written on it P6 acupressure or control group.

ps/1/2

Interviewing:

11

Each participant in both groups will be interviewed face to face to collect data related to socio-demographic status, medical and obstetrical history will be collected from both groups. Baseline data regarding frequency and severity of nausea and vomiting will be documented using (PUQE 24). Each interview will take 15 minutes.

**Implementation:** Subjects in the study group will attend scheduled small group educational and training sessions that are based on Ottawa guidelines to improve nausea and vomiting of pregnancy. The sessions will be run by the investigator as well as a licensed physiotherapist who will teach the subjects the acupressure technique. Number of subjects in each session will be 3-5. Meanwhile, subjects in the control group will be receiving the routine antenatal care, and will be equally followed up for the whole duration of the study except for the intervention.

Table (1) below shows the time, duration and contents of the educational and training sessions.

| | 1 <sup>st</sup> Session | 2 <sup>nd</sup> session |
|---|---|---|
| Time duration | For 40 minutes | For 40 minutes |
| Content | Introduction about NVP, causes, signs | Ottawa guideline (continued) |
| | and symptoms, complications and | lifestyle modifications, and the |
| | treatment. | use of acupressure by the |
| | Ottawa general guidelines for nausea | physiotherapist (how to apply |
| | and vomiting Using slides show and | pressure on the Neiguan point |

وانامرقصر

| open discussion | |
|-----------------|--------------------------------|
| . Section | of the wrist for 1 to 2 min in |
| | case of nausea). Assessment of |
| | women's ability to apply the |
| | acupressure |

After the end of the second session, Arabic booklets will be given to the intervention group to study at home. In addition, samples of recommended foods by the guidelines will be distributed to be shared by the participants during or after each session.

# Monitoring and evaluation

The study group will apply acupressure treatment by pressing for ten minutes on the anterior surface of the forearm, between the tendons of Palmaris longus and the flexor carpiradials, follow up phone calls twice a week, in addition to scheduled 2 meetings in the clinic will be done by the investigator for subjects in both study groups to assess for nausea and vomiting as well as other complaints.

# Statistical Analysis

Data analysis .Statistical Package for the Social Science (SPSS) version (20) will be used for statistical analysis of data. Collected data will be summarized and tabulated by using descriptive statistics. Inferential statistics (T-test and Chi-square) will be used to examine the differences between the study groups.P value of 0.05 will be considered as significant.

#### REFERENCES

Erick, M., Cox, J. T., andMogensen, K. M. (2018). ACOG practice bulletin 189: nausea and vomiting of pregnancy. Obstetrics and Gynecology, 131(5), 935.

ACOG Practice Bulletin No. 189: Nausea And Vomiting Of Pregnancy, Obstetrics &

Gynecology: January 2018 - Volume 131 - Issue 1 - p e15-e30 doi:

10.1097/AOG.0000000000002456

Boelig, R. C., Barton, S. J., Saccone, G., Kelly, A. J., Edwards, S. J., andBerghella, V. (2018). Interventions for treating hyperemesis gravidarum: a Cochrane systematic review and meta-analysis. The Journal of Maternal-Fetal and Neonatal Medicine, 31(18), 2492-2505.



جامعة القاهرة كلبة التمريض لجنة اخلاقيات البحث العلمي

# ثموذج موافقة مبدئية

قرار لجنة اخلاقيات البحث العلمي

اجتمعت لجنة اخلاقيات البحث العلمي بكلية التمريض - جامعة القا هرة بتاريخ ٢٦ اكتوبر ٢٠٢٠ وناقشت الملفات المقدمة من:

أسم طالبة الدكتوراه : نورا محمد الطوخي احمد قسم : تمريض صحة الام وحديثي الولادة

كلية التمريض ـ جامعة القاهرة

| رقم الدراسة: | 2020 - |
|---|---|
| اسم الدراسة<br>(باللغة الإنجليزية) | Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial) |
| اسم الدراسة<br>(باللغة العربية) | تأثير تنفيذ إرشادات "أتاوا " الغذائية على مسار الغثيان والقيئ أثناء الحمل(دراسة تجريبية عشوائية) |

اجتمعت اللجنه واطلعت على وناقشت الملفات المقدمة التالية :-

٢- ادوات البحث .

٢- الوثيقة .

١- برتوكول الدراسة .

٤- برنامج .

قرار اللجنة حيث أنها قد قامت بعمل التعديلات المطلوبة من لجنة أخلاقيات البحث العلمي المنعقدة بتاريخ ٢٦ اكتوبر 7٠٠.

هذه الموافقة صالحة لمدة سنة واحدة من تاريخ صدورها وعلى الطالبة تجديدها إذا لم تنتهى الدراسة خلال عام على الطالبة ابلاغ اللجنة عند أى تغيير أو تعديل في الملفات التي قدمت وصدر بها هذا القرار.

أعضاء اللحنة

| صوت | حضر | العضوية | الوظيفة | النوع | الاستم | م |
|---|---|---|---|---|---|---|
| ٧ | ٧ | رئيس | أستاذ متفرغ بقسم تمريض صحه الام وحديثي الولادة | أنثى | أ.د/ شادية عبد القادر حسن | 1 |
| ٧ | ٧ | عضو | أستاذ متفرغ بقسم تمريض الصحة النفسية ومدير وحدة ادارة<br>المشروعات | أنثى | أ.د/ نفيسه محمد عبد القادر | 2 |
| ٧ | ٧ | عضو | أستاذ متفرغ بقسم تمريض صحه المجتمع | أنثى | أ.د/ نجاح محمود عبده | 3 |
| ٧ | ٧ | عضو غير منتسب | استاذ متفرغ بقسم تمريض الأطفال | أنثى | أ.د/ جيهان أحمد السمان | 4 |
| ٧ | ٧ | عضو | أستاذ بكلية طب-جامعة قناة السويس وعضو الشبكة المصرية للجان أخلاقيات البحث العلمي | أنثى | أ.د/ ناهد محمد مصطفى على | 5 |
| ٧ | ٧ | مقرر | استاذ مساعد بقسم تمريض الباطني الجراحي | انثى | أ.م.د/ صفاء محمد عبد المطلب | 6 |
| ٧ | ٧ | عضو | استاذ مساعد بقسم تمريض الحالات الحرجة والطوارئ . | أنثى | أ.م.د/ فاطمة شعيب على عبد<br>الرحيم | 7 |
| ٧ | ٧ | عضو غير علمي | مسنول الشنون القانونية بالكلية | نكر | ۱. محمد ندا | 8 |
| ٧ | ٧ | عضو غير منتسب<br>وغير علمي | علاقات عامة بجامعة القاهرة | نکر | ا. حسام علاء | 9 |
| 1 | | و جر حی | | -1 | | |

عضو اللجنة (لايوجد) أحد المشرفين. أو المشاركين بالدراسة وهو عضو اللجنة حضر ولم يشارك في التصويت على القرار.

ختم اللحنة

توقيع رئيس اللجنة

المربية عبد القادر وسنوانعة مربية المربية الم

بدل فاقد

# وثيقة موافقة وإعلام بدراسة بحثية في المجال الصحي تقدم فقط للذين يوافقون على الاشتراك في هذه الدراسة

# صفحة معلومات المشارك

(رجاءا إستغرق وقتا كافيا قبل إتخاذ القرار)

:الرقم الكودي

1-عنوان البحث التأثير تنفيذ إرشادات "أتاوا" الغذائية على مسار الغثيان والقيئ أثناء الحمل (دراسة تجريبية عشوانية)" 2-الدعوة للمشاركة في الدراسة : تدعوك الباحثه للمشاركه في دراسة " إرشادات غذانية لمحاولة السيطرة على الغثيان و التقيو أثناء الحمل "

# 3 مقدمة

غثيان الحمل هو احد المتاعب البسيطة التي تحدث غالبًا خلال الشهور الأولى من الحمل. عادة ما تكون الأعراض أسوأ الشهر الثاني ، وعادة ما تتحسن في الشهر الرابع من الحمل ومع ذلك ، قد تستمر الأعراض في الشهر الثالث من الحمل وحتى الولادة، فقد تشعر النساء بالغثيان في أي وقت من اليوم، وربما تتقياً مرة أو مرتين في اليوم. عادة لا يكون ضارًا بالجنين ، على الرغم من أن القيء يوميًا له تأثير خطير على حياة المرأة مثل الفقدان الشديد للوزن، القيئ المستعصى، الجفاف، اللجوء إلى المستشفى. لذا من الافضل إتباع الإرشادات التي تساعدك على التغلب على هذا الشعور.

- وصف البحث: : تهدف هذه الدراسة إلى تقييم "تأثير إتباع إرشادات غذائية لمحاولة السيطرة على الغثيان والتقيؤ أثناء الحمل ". وسوف يتم إختيار السيدات الحوامل بعد الموافقة على الإشتراك في الدراسة. و سيتم تقديم الجلسات التعريفية للبحث وشرح الإرشادات على جلسات مختلفه مع الباحث وأخصاني العلاج الطبيعي لتعليم الضغط الإبري بالإضافة الى روتين متابعة الحمل، مع متابعة تنفيذ التعليمات.

- إستمارة جمع بيانات: سوف نحتاج منك بعض البيانات لإستكمال هذا البحث مثل بياناتك الشخصية والأجتماعيه مثل العمر، مستوى التعليم، المهنة، محل الإقامة، الوزن. بيانات خاصة بالغثيان والقيئ.

# 4- وصف تفصيلي للدراسة:-

- سيتم مقابلتك في مواعيد زيارتك لمتابعة الحمل ، و سيتم شرح هدف الدراسة لك، وسيتم جمع البيانات المتعلقة بالحالة الاجتماعية والحالة الصحية، خلال هذه المرحلة، بالإضافة إلى البيانات الأساسية المتعلقة بتكرار وشدة الغثيان والقيء. بعد الحصول على نماذج الموافقة المكتوبة.
- سيتم تحديد أيام الجلسات التدريبية وسيتم إعلامك بموعد الجلسات في اليوم السابق عبر المكالمات الهاتفية. بعد ذلك ، سيتم تقديم الإرشادات التعليمية في جلستين مدة كل منهما 60 دقيقة (3-5 حالات) في شكل محاضرة وأسئلة

وأجوبة ومناقشات جماعية (محاضرة مدتها 40 دقيقة مع عرض تقديمي للشرائح ، 20 دقيقة من الأسنلة والأجوبة ، ومناقشة المجموعة). الفاصل الزمني بين الجلسات ثلاثة أيام.

• محتوى الدورات التدريبية هو كما يلي: الجلسة الأولى ، الإرشادات التوجيهية العامة للغثيان والقيء. الجلسة الثانية ، ارشادات بخصوص تغييرات نمط الحياة ، واستخدام الطب البديل والعلاج بالضغط ويتم تدريب المشاركات بواسطة أخصانى العلاج الطبيعى، و سيتم إعطاء كتيبات للمتابعة في المنزل. خلال الأسبوع الأول من الدراسة مع متابعة الباحث لك من خلال الهاتف واللقاءات المحددة . بالإضافة إلى تلقى الرعاية الروتينية لمتابعة الحمل في المركز. إذا زاد معدل التقيو أو الجفاف لدى اى من المشاركات ، فسيتم استبعادهم من الدراسة وإحالتهم إلى المراكز الطبية لاتخاذ الإجراءات اللازمة.

# • 5 - وصف الهدف النهائي للبحث

تهدف هذه الدراسة إلى الأتى:

1. تقييم تأثير الإرشادات الغذائية لمحاولة السيطرة على الغثيان والتقيؤ أثناء الحمل.

# 6- المنافع الممكنة من الدراسة

الاشتراك بالدراسة سوف يساعد السيدات على معرفة كيفية التعامل وتخفيف المتاعب المصاحبة لغثيان وقيئ الحمل, وعدم زيادة الأعراض وتقليل اللجوء إلى دخول المستشفى بسبب تفاقم الأعراض

# 7- الأضرار التي قد تحدث

من الممكن أن تكون التعليمات غير فعالة وقد يحدث تفاقم للأعراض لديك واللجوء إلى دخول المستشفى

# 8- الإشتراك التطوعي

الإشتراك تطوعي تماما ويمكنك عدم الإشتراك أو الإنسحاب من الدراسة في أي وقت دون أن يؤثر ذلك على الخدمة الطبية المقدمة لكي في المركز.

# 9- حماية البيانات

لن يستخدم إسمك في الدراسة ، وسوف يشار إليك برمز ، وستظل هويتك غير معلنه في أي نتائج للبحث. ولن تستخدم المعلومات الخاصة بك إلا في أغراض البحث

# 10- مطومات جديدة:

سيتم إخبارك بأيه معلومات جديدة عن الدراسة .



# 11- لجنة أخلاقيات البحث العلمى:

هذا البحث تمت الموافقة عليه من قبل لجنة أخلاقيات البحث العلمي بكلية التمريض- جامعة القاهرة والتي تدفق بأن كل الشروط التي تتعلق بسلامتك وحقوقك محترمة.

وقد أعطيت الموافقة على هذا البحث بتاريخ: ....../ 2020.

#### 12- من يمكنك الإتصال به:

في حالة احتياجك لتوجيه سؤال اتصل:

اسم الباحث: نور ا محمد الطوخي أحمد

مكان العمل: كلية التمريض- جامعة القاهرة.

الهاتف: 01061001305

nouraeltoukhi @ yahoo.com:البريد الإلكتروني

إذا وافقت على الانضمام إلي هذا البحث يمكنك الأتصال برقم الهاتف السابق أو إرسال أي استفسار على البريد الإلكتروني في اي وقت إذا ما كانت لديك أسئلة أخري .

رجاءا 'استغرق وقتاً كافيا لدراسة هذه المعلومات ولا تتردد في توجيه أي أسئلة أخري للباحث في حال وجود أي غموض أو استفسارات لديك كما أن لك الحق في الاحتفاظ بنسخة من هذه الوثيقة بعد أن تقوم أنت والباحث بتوقيعها.

# قبول الإشتراك

- أعلمت بشكل صحيح بالدراسة البحثية المقترحة.
  - وضحت لي كل حقوقي بشكل واضح.
- إستلمت نسخة من وثيقة الموافقة (قبول الاشتراك).
- أوافق علي المشاركة في الدراسة المسماة:-: " تاثير تنفيذ إرشادات أوتاوا على مسار الغثيان والقيئ أثناء الحمل "
  - اشتراكك تطوعي تماماً ولديك الحق الانسحاب في أي وقت بدون إبداء تفسير أو أسياد



| | البياه | انات والمعلومات التي ستجمع نيابة عني ستكون سرية ويتم التصرف فيها طبقا لقانون حماية المعلوس |
|---|---|---|
| | الذ | تاصنة بالأشخاص وفيما يتعلق بالبيانات الشخصية. |
| • | اعلم | مت بأن البيانات المجمعة قد تستعمل في المستقبل لأي هدف علمي مع الحفاظ الكامل علي السرية. |
| | • | المنظ المنظية في مسم مس |
| | • | توقيع السيدة : التاريخ:/ |
| سم الباء | حث: | نورا محمد الطوخى أحمد |

اللقب / الوظيفة: مدرس مساعد بقسم تمريض صحة الأم وحديثي الولاده - كلية التمريض- جامعة القاهرة.

1- إعلان الرابطة العالمية والمتبني من مؤتمر الجمعية الطبية العالمية الثامن عشر الذي عقد بهلسنكي بفنلندا في يونيو 1964. والذي روجع اعوام 1975؛ 1989؛ 1989؛ 1996 وفي السادس من اكتوبر 2000 في ادنبرة اسكتلندا www.wma.net

التاريخ :..... /.....

- 2- توجيهات ICH-GCP للممارسة السريرية الجيدة CPMB/ICH/35/95 سبتمبر 1997.
- 3- التوجيهات الأخلاقية العالمية للبحث الطبي الحيوي المتضمن آدميين ، مجلس المنظمات العالمية للعلوم الطبية
   3- التوجيهات الأخلاقية العالمية للبحث الطبي الحيوي المتضمن آدميين ، مجلس المنظمات العالمية للعلوم الطبية
  - 4- الصحة العالمية: الترجيهات العلمية للجنة الأخلاقية لمراجعة البحوث الطبية الحيوية، جنيف 2000.

# وثيقة موافقة وإعلام بدراسة بحثية في المجال الصحى تقدم فقط للذين يوافقون على الاشتراك في هذه الدراسة مرادمات المشاد الدرجم عق 2

# صفحة معلومات المشارك (مجموعة 2)

(رجاءا إستغرق وقتا كافيا قبل إتخاذ القرار)

#### :الرقم الكودي

1-عنوان البحث " تأثير تنفيذ إرشادات "أتاوا " الغذانية على مسار الغثيان والقيئ أثناء الحمل (دراسة تجريبية عشوانية)" 
2-الدعوة للمشاركة في الدراسة : تدعوك الباحثه للمشاركه في دراسة " إرشادات غذانية لمحاولة السيطرة على الغثيان والتقيؤ أثناء الحمل "

# 3 مقدمة

غثيان الحمل هو احد المتاعب البسيطة التي تحدث غالبًا خلال الشهور الأولى من الحمل. عادة ما تكون الأعراض أسوأ الشهر الثاني ، وعادة ما تتحسن في الشهر الرابع من الحمل. ومع ذلك ، قد تستمر الأعراض في الشهر الثالث من الحمل وحتى الولادة، فقد تشعر النساء بالغثيان في أي وقت من اليوم، وربما نتقياً مرة أو مرتين في اليوم. عادة لا يكون ضارًا بالجنين ، على الرغم من أن القيء يوميًا له تأثير خطير على حياة المرأة، مثل الفقدان الشديد للوزن، القيئ المستعصى، الجفاف، اللجوء الى المستشفى. لذا من الافضل إتباع الإرشادات التي تساعدك على التغلب على هذا الشعور.

- وصف البحث: تهدف هذه الدراسة إلى تقييم "تأثير إتباع إرشادات غذانية لمحاولة السيطرة على الغثيان والتقيؤ أثناء الحمل ". وسوف يتم إختيار السيدات الحوامل بعد الموافقة على الإشتراك في الدراسة. و سيتم تقديم الجلسات التعريفية للبحث وشرح الإرشادات على جلسات مختلفه مع الباحث بالإضافة الى روتين متابعة الحمل.

-إستمارة جمع بيانات: سوف نحتاج منك بعض البيانات لإستكمال هذا البحث مثل بياناتك الشخصية والأجتماعيه مثل العمر، مستوى التعليم، المهنة، محل الإقامة، الوزن. بيانات خاصة بالغثيان والقيئ.

# 4- وصف تفصيلي للدراسة:-

- سيتم مقابلتك في مواعيد زيارتك لمتابعة الحمل ، و سيتم شرح هدف الدراسة لك، وسيتم جمع البيانات المتعلقة بالحالة الاجتماعية والحالة الصحية، خلال هذه المرحلة، بالإضافة إلى البيانات الأساسية المتعلقة بتكرار وشدة الغثيان والقيء.
   بعد الحصول على نماذج الموافقة المكتوبة ،
  - سيتم تحديد أيام للجلسات وسيتم إعلامك بموعد الجلسات في اليوم السابق عبر المكالمات الهاتفية.

# 5 - وصف الهدف النهائي للبحث

تهدف هذه الدراسة إلى الأتى:



تهدف هذه الدراسة إلى الأتى:

تقييم تأثير الإرشادات الغذائية لمحاولة السيطرة على الغثيان والتقيؤ أثناء الحمل.

### 6- المنافع الممكنة من الدراسة

الاشتراك بالدراسة سوف يساعد السيدات على معرفة كيفية التعامل وتخفيف المتاعب المصاحبة لغثيان وقيئ الحمل, وعدم زيادة الأعراض وتقليل اللجوء إلى دخول المستشفى بسبب تفاقم الأعراض

# 7- الأضرار التي قد تحدث

من الممكن أن تكون التعليمات غير فعالة وقد يحدث تفاقم للأعراض لديك واللجوء إلى دخول المستشفى

#### 8- الإشتراك التطوعي

الإشتراك تطوعي تماما ويمكنك عدم الإشتراك أو الإنسحاب من الدراسة في أي وقت دون أن يؤثر ذلك علي الخدمة الطبية المقدمة لكي في المركز.

#### 9- حماية البيانات

لن يستخدم إسمك في الدراسة ، وسوف يشار إليك برمز ، وستظل هويتك غير معلنه في أي نتائج للبحث. ولن تستخدم المعلومات الخاصة بك إلا في أغراض البحث

#### 10- مطومات جديدة:

سيتم إخبارك بأيه معلومات جديدة عن الدراسة .

#### 11- لجنة أخلاقيات البحث العلمى:

هذا البحث تمت الموافقة عليه من قبل لجنة أخلاقيات البحث العلمي بكلية التمريض- جامعة القاهرة والتي تدقق بأن كل الشروط التي تتعلق بسلامتك وحقوقك محترمة.

وقد أعطيت الموافقة على هذا البحث بتاريخ: ....../....../ 2020.

#### 12- من يمكنك الإتصال به:

في حالة احتياجك لتوجيه سؤال اتصل:

اسم الباحث: نورا محمد الطوخي أحمد



مكان العمل: كلية التمريض- جامعة القاهرة.

الهاتف: 01061001305

nouraeltoukhi @ yahoo.com:البريد الإلكتروني

إذا وافقت على الانضمام إلى هذا البحث يمكنك الأتصال برقم الهاتف السابق أو إرسال أي استفسار على البريد الإلكتروني في اى وقت إذا ما كانت لديك أسئلة أخري .

رجاءا 'استغرق وقتاً كافيا لدراسة هذه المعلومات ولا تتردد في توجيه أي أسئلة أخري للباحث في حال وجود أي غموض أو استفسارات لديك كما أن لك الحق في الاحتفاظ بنسخة من هذه الوثيقة بعد أن تقوم أنت والباحث بتوقيعها.

## قبسول الإشتسراك

- أعلمت بشكل صحيح بالدراسة البحثية المقترحة.
  - وضحت لى كل حقوقى بشكل واضح.
- إستلمت نسخة من وثيقة الموافقة (قبول الاشتراك).
- أوافق علي المشاركة في الدراسة المسماة:-: " تاثير تنفيذ إرشادات أوتاوا على مسار الغثيان والقيئ أثناء
  - اشتراكك تطوعى تماماً ولديك الحق الانسحاب في أي وقت بدون إبداء تفسير أوأسباب.
- البيانات والمعلومات التي ستجمع نيابة عني ستكون سرية ويتم التصرف فيها طبقا لقانون حماية المعلومات الخاصة بالأشخاص وفيما يتعلق بالبيانات الشخصية.
  - أعلمت بأن البيانات المجمعة قد تستعمل في المستقبل لأي هدف علمي مع الحفاظ الكامل على السرية.

| • اسم السيدة: |
|---|
| <ul> <li>توقیع السیدة :</li> <li>التاریخ:/</li> </ul> |
| اسم الباحث: نورا محمد الطوخى أحمد |
| اللقب / الوظيفة: مدرس مساعد بقسم تمريض صحة الأم وحديثي الولاده - كلية التمريض- جامعة القاهرة. |
| توقيع الباحث : التاريخ : التاريخ الباحث : التاريخ السادة التاريخ التا |
| عليّ المريف عليه المريف عليه المريف عليه المريف عليه المريف المري |

# هذه الوثيقة أعدت مع الأخذ في الاعتبار لكلا من:

- إعلان الرابطة العالمية والمتبنى من مؤتمر الجمعية الطبية العالمية الثامن عشر الذي عقد بهلسنكي بفنلندا في يونيو 1964 والذي روجع اعوام 1975؛ 1983؛ 1989؛ 1996 وفي السادس من اكتوبر 2000 في ادنيرة السكتلندا www.wma.net
  - 2- توجيهات ICH-GCP للممارسة السريرية الجيدة CPMB/ICH/35/95 سبتمبر 1997.
- 3- التوجيهات الأخلاقية العالمية للبحث الطبي الحيوي المتضمن أدميين ، مجلس المنظمات العالمية للعلوم الطبية
   (CIOMS)، جنيف عام 1993.
  - الصحة العالمية: التوجيهات العلمية للجنة الأخلاقية لمراجعة البحوث الطبية الحيوية، جنيف 2000.





جاسعة القاهرة كلبة التعريض لجنّة لفلاقيات البحث العلمي

# نموذج موافقة نهائية

قرار لجنة أخلاقيات البحث العلمى

اجتمعت لجنة اخلاقيات البحث العلمي بكلية التمريض - جامعة القاهرة بتاريخ ١٨ اكتوبر ٢٠٢١ وناقشت الملفات المقدمة من:

أسم طالبة الدكتوراه: نورا محمد الطوخي احمد قسم: تمريض صحة الام وحديثي الولادة

كلية التمريض - جامعة القاهرة

| 2020 - | رقع الدارسة : |
|---|---|
| Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial) | اسم الدارسة<br>(باللغة الإنجليزية) |
| تأثير تنفيذُ إرشادات "أتاوا " الغذائية على مسار الغثيان والقيئ أثناء الحمل(دراسة تجريبية عشوائية) | اسم الدازمية<br>(باللغة العربية) |

| تم مراجعة استمارة قبول الاشتراك المعتمدة من لجنة اخلاقيات البحث العلمي بكلية التمريض - جامعة القاهرة | قرار اللجنة |
|---|---|
| الخاصه بطالبة الدكتوراه: نورا محمد الطوخى على التي جمع بها البيانات الخاصه برساله الدكتوراه، وبناءا | فراز اللجنة |
| عليه يمنح الموافقة النهائية على ذلك. | 1 |

أعضاء اللجنة

| صوت | حضر | العضوية | الوظيفة | النوع | الاسم | م |
|---|---|---|---|---|---|---|
| ٧ | ٧ | رنیس | أستاذ متفرغ بقسم تمريض صحه الام وحديثى الولادة | أنثى | أ.د/ شادية عبد القادر حسن | 1 |
| ٧ | ٧ | عضو | أستاذ متفرغ بقسم تمريض الصحة النفسية ومدير وحدة ادارة المشروعات | أنثى | أد/ نفيسه محمد عبد القادر | 2 |
| ٧ | ٧ | عضو | أستاذ متفرغ بقسم تمريض صحه المجتمع | أنثى | أ.د/ نجاح محمود عبده | 3 |
| ٧ | ٧ | عضو غير منتسب | استاذ متفرغ بالمعهد القومى للاورام | | أ.د/ عاطف بدران | 4 |
| ٧ | ٧ | مقرر | أستاذ متفرغ بقسم تمريض الأطفال | أنثى | أ.د/ جيهان أحمد السمان | 5 |
| ٧ | ٧ | عضو | أستاذ بكلية طب جامعة قناة السويس وعضو الشبكة المصرية للجان أخلاقيات البحث العلمي | أنثى | أد/ ناهد محمد مصطفى على | 6 |
| ٧ | ٧ | عضو | استاذ مساعد بقسم ادارة التمريض . | أنثى | أ.م.د/ سحر حسن على البنان | 7 |
| ٧ | ٧ | عضو | استاذ مساعد بقسم تمريض الباطني الجراحي . | أنثى | أ.م.د/ داليا صلاح الدين عبد المنعم<br>السعداوي | 8 |
| ٧ | ٧ | عضو غير علمي | مسنول الشنون القانونية بالكلية | نكر | ا. أحمد محمود محمود حسن | 9 |
| ٧ | ٧ | عضو غیر منتسب<br>وغیر علمی | اخصائي موارد بشرية ثالث بكلية طب الفم والاسنان | ذكر | ١. ابراهيم عبد الباقى عبد الحميد | 10 |

عضو اللجنة (لا يوجد) أحد المشرفين. أو المشاركين بالدراسة وهو عضو اللجنة حضر ولم يشارك في التصويت على القرار.

توقيع رئيس اللجنة के निय ह

أستاذ متفرغ بقسم تمريض صحه الام وحديثي الولادة

كلية التمريض - جامعة القاهرة - المنيل - داخل حرم مستشفيات القصر العيني (المبنى الاكاديمي الدور الثالث)



IORG0006883 Cairo University

RHDIRB2019041701 FWA 00026458 valid to 22-01-2023

# Model final approval

**Decision of the Scientific Research Ethics Committee** 

The Scientific Research Ethics Committee met at the Faculty of Nursing - Cairo University on October 18, 2021 and discussed the files submitted by:

Postgraduate Student Name: Noura Mohamed Eltoukhi

Department: Obstetric and newborn health nursing- Faculty of Nursing - Cairo University

| Study number: | 2020 - 44 |
|---|---|
| Study name<br>(In English) | Effect of Implementing Ottawa Nutritional Guidelines on the Course of Nausea and Vomiting During Pregnancy (A Randomized Control Trial) |

| decision | The application form approved by the Scientific Research Ethics Committee at the Faculty of Nursing - Cairo University has been reviewed for the Mrs. Noura Mohamed Eltoukhi which he collected his scientific doctorate thesis data, and accordingly, the final approval is granted. |
|---|---|
|---|---|

| | Committee members | | | Attendance | Opinion |
|---|---|---|---|---|---|
| No. | Name | Occupation | Affiliation | Attendance | Opinion |
| 1. | Prof. Shadia Abdel Qader Hassan | Professor Emeritus of Maternal and<br>Newborn Health Nursing | Chairman<br>of the<br>Committee | ٧ | ٧ |
| 2. | Prof. Nafisa Mohamed Abdel Qader | Professor Emeritus in the Department<br>of Mental Health Nursing and Director<br>of the Project Management Unit | Committee<br>member | ٧ | ٧ |
| 3. | Prof. Najah Mahmoud Abdo | Emeritus Professor, Department of<br>Community Health Nursing | Committee<br>member | ٧ | ٧ |
| 4. | Prof. Atef Badran | Emeritus Professor at the National<br>Cancer Institute | Committee<br>member | ٧ | ٧ |
| 5. | Prof. Gihan Ahmed Al-Samman | Professor Emeritus of Pediatric<br>Nursing | Committee<br>member | ٧ | ٧ |
| 6. | Prof Nahed Muhammad Mustafa Ali | Professor at the Faculty of Medicine -<br>Suez Canal University and a member of<br>the Egyptian Network of Scientific<br>Research Ethics Committees | Committee<br>member | ٧ | ٧ |
| 7. | Ass.prof. Sahar Hassan Ali Banan | Assistant Professor, Department of Nursing Administration. | Committee<br>member | ٧ | ٧ |
| 8. | Ass.prof. Dalia Salah El Din Abdel<br>Moneim El Saadawy | Assistant Professor, Department of<br>Surgical Internal Nursing. | Commission decision | ٧ | ٧ |
| 9. | Mr. Ahmed Mahmoud Mahmoud<br>Hassan | College legal affairs officer | Committee<br>member | ٧ | ٧ |
| 10. | Mr. Ibrahim Abdel Baqi Abdel Hamid | Third HR Specialist, Faculty of Oral and Dental Medicine | Committee<br>member | ٧ | ٧ |

Committee member (no) one of the supervisors. Or the study participants who is a member of the committee who attended and participated in voting on the decision.

Chairman's signature

Prof. Shadia A. Hassan

Professor of Materna.lNewborn Health Nursing-Faculty of Nursing - Cairo University

Hanan Falmy 24-9-2023